CLINICAL TRIAL: NCT00083395
Title: Utility of Isoproterenol Challenge Test to Detect Disease in Patients With Incomplete Diagnostic Criteria for Arrhythmogenic Right Ventricular Cardiomyopathy
Brief Title: Isoproterenol Challenge to Detect Arrhythmogenic Right Ventricular Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040194; 04-CC-0194
Record Dates: First submitted 2004-05-22; First posted 2004-05-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-12

CONDITIONS: Arrhythmic Right Ventricular Cardiomyopathy
Keywords: ARVC/ARVD; Genetics; Sudden Death; Heart; MRI; Cardiomyopathy; Arrhythmogenic Right Ventricular; ARVC; Healthy Volunteer; HV
MeSH Terms: conditions — Death, Sudden; Cardiomyopathies

SUMMARY:
This study will examine the usefulness of a new test called an isoproterenol challenge in patients with arrhythmogenic right ventricular cardiomyopathy (ARVC) and family members who may have the disease but do not have clear-cut evidence of it. ARVC is a rare condition that runs in families. Heart muscle is replaced with fatty, scar-like tissue, especially in the right ventricle (lower pumping chamber of the heart), and can sometimes extend to the left ventricle (the main pumping chamber). The fat can interfere with the heartbeat, producing abnormal heart rhythms, such as ventricular tachycardia (VT) - a very fast heartbeat that can cause sudden death, especially in young people. Isoproterenol is a drug that increases heart rate and heart muscle contractions. In isoproterenol challenge, subjects are given increasing doses of the drug through a catheter (see details below) to try to produce an abnormal heart rhythm.

ARVC is hard to diagnose with current tests. This study will see if isoproterenol challenge provokes VT in patients with the disease and can confirm the diagnosis; if it can detect the disease in family members better than currently available tests; and if it provokes abnormal rhythms in healthy control subjects. In addition, the study will explore the genetics of ARVC and determine whether infection could contribute to its development.

Patients with ARVC, their family members, and normal volunteers 18 years of age and older may be eligible for this study. Candidates are screened with a medical history and physical examination, electrocardiogram (EKG), treadmill and bicycle exercise testing, and an echocardiogram (ultrasound test of the heart).

Participants undergo the following tests and procedures:

* Blood tests - Blood is collected to study the genetics of ARVC, to test for evidence of old infections, and to measure brain natriuretic peptide - a hormone that can increase with development of heart failure.
* Heart magnetic resonance imaging (MRI). This test looks at heart structure and function. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. The subject lies on a table that is moved into the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking sounds that occur during the scanning process. At some time during the test, the subject is given a contrast agent called gadolinium through a catheter (thin, flexible tube) in a vein to improve the scan pictures. The scan time varies from 30 to 90 minutes, with most scans lasting 60 minutes. (Control subjects do not undergo MRI.)
* Isoproterenol challenge. Subjects are given increasing doses of isoproterenol through a catheter until the heart rate reaches 100 to 120 beats per minute for no more than 1 hour. A special EKG records heart rhythm during the test and an echocardiogram records right and left ventricular function.
* QRST surface mapping EKG. This special EKG, done with 64 or 120 leads, maps abnormalities of heart rhythm and cardiac conduction during the isoproterenol challenge. These tests are like a regular EKG, except that more leads are placed on the chest, and on the back as well.

Patients and family members who wish to have follow-up visits may return to the NIH Clinical Center once a year for 5 years for guidance about therapy based on clinical considerations and new information or investigations.

DETAILED DESCRIPTION:
Arrhythmogenic right ventricular cardiomyopathy (ARVC) formerly referred to as arrhythmogenic right ventricular dysplasia (ARVD) is a familial hetergenous clinical and molecular disease characterized by dilatation and dysfunction of the right ventricle and ventricular arrhythmias. The ventricular arrhythmias are heart rate and catecholamine dependent. Not infrequently, there is involvement of the left ventricle. The diagnosis of ARVC is critical as therapy including implantable defibrillators may prevent sudden death. However, identification of affected family members remains a major challenge due to limitation of current imaging and diagnostic techniques. We propose (1) to establish the sensitivity and specificity of the isoproterenol challenge test for ARVC by testing both patients with known ARVC and healthy volunteers; (2) to estimate the proportion of family members who present with incomplete criteria for ARVC but are subsequently diagnosed with the condition by an isoproterenol challenge test; and, (3) to study the inheritance of ARVC and the potential role of occult infection in its development.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with ARVC:

Either gender, aged greater than 5 years.

The presence of two major criteria; one major and two minor criteria; or four minor criteria from separate diagnostic categories.

Normal Volunteers:

Age and gender matched with ARVC patients, age greater than 18 years.

No known cardiac disease.

Normal EKG, normal echocardiogram, normal Bruce protocol treadmill exercise test.

Family Members of Patients with ARVC:

Either gender, aged greater than 5 years.

A proband with ARVC

EXCLUSION CRITERIA:

Patients with ARVC:

Pregnancy or lactation excludes tests with potential risk, e.g. radiation, isoprenaline, MRI, but does not exclude 12-lead ECG and echocardiogram.

Coronary artery disease.

Known infiltrate or congenital heart disease that could mimic the appearances of ARVC.

Asthma prevents participation in Isoproterenol infusion.

Any other condition that would prevent participation in the study.

Normal Volunteers:

Pregnancy or lactation.

Asthma.

Coronary artery disease, hypertension, diabetes, hypertrophic cardiomyopathy, or other known cardiomyopathy.

Known infiltrative or congenital heart disease that could mimic the appearances of ARVC.

Any Acute or chronic illness.

Chronic drug therapy.

Family Members of Patients with ARVC:

Pregnancy or lactation excludes tests with potential risk, e.g. radiation, isoprenaline, MRI, but does not exclude 12-lead ECG and echocardiogram.

Coronary artery disease.

Known infiltrative or congenital heart disease that could mimic the appearances of ARVC.

Asthma prevents participation in Isoproterenol infusion.

Any other condition that would prevent participation in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2004-05; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] DALLA VOLTA S, BATTAGLIA G, ZERBINI E. "Auricularization' of right ventricular pressure curve. Am Heart J. 1961 Jan;61:25-33. doi: 10.1016/0002-8703(61)90513-0. No abstract available. PMID 13719440
- [Background] Basso C, Thiene G, Nava A, Dalla Volta S. Arrhythmogenic right ventricular cardiomyopathy: a survey of the investigations at the University of Padua. Clin Cardiol. 1997 Apr;20(4):333-6. doi: 10.1002/clc.4960200406. PMID 9098590
- [Background] Marcus FI, Fontaine GH, Guiraudon G, Frank R, Laurenceau JL, Malergue C, Grosgogeat Y. Right ventricular dysplasia: a report of 24 adult cases. Circulation. 1982 Feb;65(2):384-98. doi: 10.1161/01.cir.65.2.384. PMID 7053899